CLINICAL TRIAL: NCT01775436
Title: Palliative Care in People Living With HIV/AIDS: Integrating Into Standard of Care
Acronym: FACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Georgetown University (Other); George Washington University (Other); VA Medical Center (Unknown); Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Maureen Lyon, Principal Investigator, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01NR01405201
Record Dates: First submitted 2012-12-20; First posted 2013-01-25 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2019-03

CONDITIONS: HIV
Keywords: palliative care; HIV/AIDS; quality of life; adherence; spiritual; threat appraisal; treatment congruence; treatment preferences; dialysis; hospitalization; communication; family intervention; Family Centered Advance Care Planning; decision making; advance care planning; end of life
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Communication; Death

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor did not know which study arm the participant was randomized to.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Living Control (Active Comparator): Two-60 to 90 minute sessions scheduled one week apart.
  Session 1: Developmental History: Goal: To take a non-medical developmental history. The Research Assistant (RA)-Control will conduct the session in a structured interview format. Administered with all medical questions removed to prevent any risk of contamination with the experimental condition.
  Session 2: Nutrition and Exercise: Assess nutritional status and provide advice for maintaining optimal nutrition to boost immune functioning. Administered by the RA Control and will be videotaped to control for what occurs in the FACE intervention.
  Interventions: Behavioral: FAmily-CEntered Advance Care Planning; Behavioral: Healthy Living Control
- FAmily-CEntered Advance Care Planning (Experimental): Two-60 to 90 minute sessions scheduled one week apart.
  Session 1: Respecting Choices Interview (R)to facilitate conversations and shared decision-making between the patient and surrogate about palliative care & prepare the surrogate to be able to fully represent the patient's wishes.
  Session 2: Five Wishes (C). Patient selects which person the patient wants to make health care decisions for him/her; the kind of medical treatment the patient wants; how comfortable the patient wants to be; how the patient wants people to treat him/her; what patient wants loved ones to know; and any spiritual or religious concerns the patient may have.
  Interventions: Behavioral: FAmily-CEntered Advance Care Planning; Behavioral: Healthy Living Control

INTERVENTIONS:
Behavioral: FAmily-CEntered Advance Care Planning — Two-60 to 90 minute sessions scheduled one week apart.
  Session 1: Respecting Choices Interview (R)to facilitate conversations and shared decision-making between the patient and surrogate about palliative care & prepare the surrogate to be able to fully represent the patient's wishes.
  Session 2: Five Wishes (C). Patient selects which person the patient wants to make health care decisions for him/her; the kind of medical treatment the patient wants; how comfortable the patient wants to be; how the patient wants people to treat him/her; what patient wants loved ones to know; and any spiritual or religious concerns the patient may have.
  Other Names: FACE
Behavioral: Healthy Living Control — Session 1: Developmental History: Goal: To take a non-medical developmental history. The RA-Control will conduct the session in a structured interview format. Administered with all medical questions removed to prevent any risk of contamination with the experimental condition.
  Session 2: Nutrition and Exercise: Assess nutritional status and provide advice for maintaining optimal nutrition to boost immune functioning. Administered by the RA Control and will be videotaped to control for what occurs in the FACE intervention.
  Other Names: HLC

SUMMARY:
Our goal is to advance palliative care with persons living with AIDS (PLWA) or life-limiting co-morbidities to decrease suffering and increase quality of life (QOL). Left without advance care planning (ACP) for end-of-life decision, miscommunication and disagreements may result in families being charged with neglect or court battles over treatment choices, unmet care or delivery of unnecessary or unwanted care, and non-relative caregivers being dismissed (e.g. gay partners). We hope to increase families' understandings of their family member's wishes for end-of-life care to decrease conflict through the FAmily-CEntered Advance (FACE) Care Planning intervention. We will also study communication, quality of life, and spiritual struggle. Families will be randomized into either the Control (N=96 families) or the FACE Intervention (n=192 dyads). FACE families will meet with a trained/certified researcher for two 60-minute sessions scheduled one week apart: Session 1: The Respecting Choices Interview®; and Session 2: Completion of The Five Wishes©. Control families will also meet with a researcher for two 60-minute sessions scheduled one week apart: Session 1: Developmental History; and Session 2: Nutrition and Exercise. Questionnaires will be administered five times, Baseline and at 3, 6, 12 and 18 month post-intervention, for an average of 2 years.

AIM 1. To determine the efficacy of FACE on congruence in treatment preferences between PLWA and their surrogates over time, and the effect of the pattern of congruence development trajectory on healthcare utilization (i.e., distal outcomes: number of hospitalizations, dialysis, ER visits).

Hypothesis A: Development of congruence may not be homogeneous and FACE may influence the pattern of congruence development.

Hypothesis B: Different patterns of congruence development may have different effects on health care utilization.

Hypothesis C: Compared to Controls, FACE participants will better maintain congruence over time.

AIM 2. To determine the efficacy of FACE on key components of QOL for PLWA. Hypothesis: FACE participants will increase or better maintain psychosocial QOL compared to Controls.

AIM 3. To minimize health disparities in ACP between Blacks and non Blacks and identify factors associated with disparities.

Hypothesis: Blacks in the FACE intervention will complete advance directives at a rate comparable to non Blacks, and at significantly greater rates compared to Controls.

DETAILED DESCRIPTION:
Our goal is to advance palliative care with persons living with AIDS (PLWA) or life-limiting co-morbidities aimed at relieving suffering and maximizing quality of life. One objective is to identify variables which influence decision-making with respect to advance care planning (ACP) for PLWA, as well as to determine the unique person-centered needs of subgroups of PLWA, as these are unknown. The negative consequences of no ACP or poor ACP include: unmet care or delivery of unnecessary or unwanted care, conflict erupting in the ICU, or the importance of non-relative caregivers being dismissed, for example gay partners. A second objective is to identify a "best approach" for standard of care in ACP, a key component of palliative care, as an end of life support. This approach may minimize health disparities in the likelihood of both identifying a surrogate decision-maker and using advance directives. We propose building on our evidence based, theoretical model, FAmily-CEntered (FACE) Advance Care Planning intervention, an HIV specific ACP program for Black teens which gained acceptance and demonstrated efficacy through increased congruence in treatment preferences and universal complete of advance directives with a surrogate decision-maker. Given the demonstrated needs and benefits of ACP and the low utilization among adult Black PLWA, we propose meeting this need by building on our FACE model with adults living with advanced AIDS and/or life-limiting co-morbidities in Washington, District of Columbia (DC) a city with endemic HIV and significant health disparities in death rates by race in an adequately-powered, randomized, clinical, 2-arm, single-blinded, controlled trial. We will test the efficacy of the FACE intervention for increasing congruence in end-of-life treatment preferences between PLWA and their surrogate decision-maker, to determine if increased congruence can be maintained over time. We will also determine if FACE is acceptable to primarily Black inner city adult PLWA. We will recruit from four hospital-based clinics and randomize 288 patient/surrogate dyads (N=576 subjects) in a 2:1 ratio to either FACE Intervention (N=192 dyads) or Control (N=96 dyads). Participants with HIV dementia, suicidality, homicidality or psychosis will be excluded. Two 60-minuted sessions will be conducted with a trained/certified facilitator at weekly intervals: FACE Session 1: The Respecting Choices Interview (R); Session 2: Completion of The Five Wishes (c). Control will also be administered in a dyadic format: Session 1: Developmental History; Session 2: Nutrition and Exercise. Standardized self-report measures will be administered at baseline, 3 month post-intervention 6 month post-intervention, 12 month post-intervention, and 18 month post-intervention. Thus, participants will be followed for an average of 2 years. This will be the first study to test an ACP model, integrating person-centered (GMM) and variable-centered analysis (GEE) to assess study outcomes.

ELIGIBILITY:
Patient Inclusion Criteria:

* HIV positive outpatients or inpatients with detectable viral load (>200 copies) twice in the past 1 year period OR CD4 count <200 OR with a co-morbidity that may significantly limit life expectancy, including malignancy, cirrhosis, cardiomyopathy, etc.
* Patients with AIDS receiving dialysis, inpatients or outpatients
* Patients not in the Intensive Care Unit (ICU)
* Age 21 years or older
* All ethnic groups
* Male or female
* Knows his/her HIV status
* English speaking
* Absence of active psychosis or homicidal or suicidal ideation, determined at baseline screening by a trained research assistant as assessed by questions from a structured questionnaire
* Absence of HIV dementia, determined at screening using the HIV Dementia Scale cut off score of <10
* No evidence of developmental delay
* Consent from surrogate
* Consent from persons living with AIDS (PLWA) aged 21 or older

Surrogate Decision-maker inclusion criteria:

* Selected by patient
* Age 18 or older
* Willingness to discuss problems related to HIV and End Of Life (EOL)
* Absence of active psychosis, homicidal ideation, or suicidal ideation determined at baseline screening by trained RA
* Absence of HIV dementia, determined at screening using the HIV Dementia Scale cut off score of <10
* English speaking
* Consent to participate
* Knows HIV status of patient

Patient Exclusion Criteria:

* Patients in the ICU
* Age under 21 years old
* Patient unaware of HIV status
* Active psychosis or homicidal or suicidal ideation, determined at baseline screening by a trained research assistant as assessed by questions from a structured questionnaire
* Presence fo HIV Dementia at baseline
* Developmental delay
* Unable to find willing consented surrogate

Surrogate Decision-maker Exclusion Criteria:

* Surrogate under age of 18 years old
* Unwilling to discuss problems related to HIV and EOL
* Active psychosis or homicidal or suicidal ideation, determined at baseline screening by a trained research assistant as assessed by questions from a structured questionnaire
* Not an English speaker
* Unwilling to consent to participate and does not know HIV status of patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2013-10-13 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Statement of Treatment Preferences | Baseline and 3, 6, 12, 18 month post-intervention
  Measured by the Statement of Treatment Preferences. This measure was adapted using experts and community advisory board. It is a tool to express values and goals related to future medical decisions regarding frequently occurring situations specific to HIV/AIDS.Multiple Time Frames are needed as the Primary Outcome measure is going to report a change over time, per Aim 1: "to sustain congruence in treatment preferences between PLWA and their surrogate over time" compared to controls.

SECONDARY OUTCOMES:
Lyon Advance Care Planning Survey (Patient and Surrogate Version) | at baseline
  A 31-item instrument that assesses palliative care needs of PLWA of Black and non Black PLWA in DC metropolitan area
Palliative Care Outcome Scale (POS) | Baseline, and 3, 6, 12 and 18 month post-intervention
  This scale is a valid and reliable measure of patient's current health, social and psychological status.We are conducting a longitudinal study and therefore looking at multiple time frames for change in palliative care over time.
Medical Outcomes Study-HIV (MOS-HIV) | Baseline, and 3, 6, 12 and 18 month post-intervention
  Measures HIV specific Health Related Quality of Life; general health perceptions; pain; physical, role, cognitive and social functioning; mental health; energy/fatigue; health distress and quality of life. This is a longitudinal study requiring multiple time frames so we can report change in quality of life over time, related to HIV specific symptoms.

OTHER OUTCOMES:
HIV Dementia Scale | Screen for eligibility at Baseline, 3, 6, 12 and 18 months post intervention
  Rapid screener to identify HIV dementia, which is an exclusion criteria. However, once enrolled in the study we will track changes in status over time, per the longitudinal nature of this study.
Psychological Interview | Baseline to screen to determine eligibility
  Questions to screen for homicidality and psychosis
Patient Health Questionnaire (PHQ-9) | Baseline screening to determine if eligible for participation, then at 3, 6, 12 and 18 month post-intervention follow-up
  Patients or surrogates who present with severe depression or suicidality are excluded from this study. However, once enrolled levels of depressive symptoms will be monitored over the course of this longitudinal study.
Medication Adherence Self Report Inventory (MASRI) | Baseline and 3, 6, 12 and 18 month follow-up
  Validated self-report measure of medication adherence, using the Visual Analogue Scale for estimated adherence in the past month. Measured multiple times as part of this longitudinal study.
Brief Multidimensional Measurement of Religiousness/Spirituality (BMMRS-adapted) | Baseline and 3, 6, 12 and 18-month post intervention
  Assesses the construct of spiritual functioning, specifically subscales for Forgiveness, Values and Believes will be used for study purposes.
Brief Religious Coping Questionnaire (Brief RCOPE) | Baseline and 3, 6, 12 and 18-month post-intervention
  Assesses positive and negative religious coping methods. Study will use 14-item version.
Satisfaction Scale | Immediately following Session 1 and Session 2, week 2 and week 3 of the study
  Process measure developed in pilot study to assess satisfaction.
Longitudinal Satisfaction Questionnaire | 3, 6, 12 and 18 month post-intervention
  Process measure to assess longitudinal satisfaction with future decision making.
Medical Chart Abstraction | Baseline and 3, 6, 12 and 18 month post intervention
  Mode of transmission, Cluster of Differentiation 4 (CD4) count, viral load, hospitalization, emergency room visit or dialysis since last study visit.
Threat Appraisal Scale (TAS) | Baseline, 3, 6, 12 and 18 month post-intervention
  Threat Appraisal Scale (TAS)is a questionnaire administered to the adolescent during baseline assessment only. This measure will retrospectively estimate the adolescent's threat appraisal of cancer when adolescent learned of cancer diagnosis. Test-retest reliability for this measure ranges from .68 in younger children to .93 in older children. TAS scores are found to demonstrate a high degree of agreement with children's open-ended descriptions of negative life events, indicating adequate convergent validity of this measure. Theoretically, threat appraisal is related to Lazarus' concept of primary appraisal, particularly to the way in which the event threatens the child's commitments, goals, or values. Higher threat appraisals should lead to negative arousal and coping and to increased psychological symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E Lyon, PhD, Principal Investigator — Children's National Research Institute
Locations (5):
- United States (5):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Institute for Clinical Research, Inc. (Affiliated with Department of Veterans Affairs Medical Center of Washington, DC), Washington D.C., District of Columbia
  - MedStar Health Research Institute/Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make de-identified individual participant data (IPD) collected in this study, which are not part of the specific aims, available for secondary analysis, to be shared with other researchers by submitting a request to the PI, Dr. Lyon.
Supporting Information: Study Protocol
Time Frame: Data will become available on June 30, 2018 and for a period of two years.
Access Criteria: Researchers or graduate students in need of a master's theses or dissertation project from academic settings, e.g. university or academic/research hospital will be allowed to have access to de-identified data.
  Contact the PI Dr. Lyon at mlyon@childrensnational.org.

REFERENCES:
- [Result] Kimmel AL, Wang J, Scott RK, Briggs L, Lyon ME. FAmily CEntered (FACE) advance care planning: Study design and methods for a patient-centered communication and decision-making intervention for patients with HIV/AIDS and their surrogate decision-makers. Contemp Clin Trials. 2015 Jul;43:172-8. doi: 10.1016/j.cct.2015.06.003. Epub 2015 Jun 2. PMID 26044463
- [Result] Lyon ME, Squires L, D'Angelo LJ, Benator D, Scott RK, Greenberg IH, Tanjutco P, Turner MM, Weixel TE, Cheng YI, Wang J. FAmily-CEntered (FACE) Advance Care Planning Among African-American and Non-African-American Adults Living With HIV in Washington, DC: A Randomized Controlled Trial to Increase Documentation and Health Equity. J Pain Symptom Manage. 2019 Mar;57(3):607-616. doi: 10.1016/j.jpainsymman.2018.11.014. Epub 2018 Nov 23. PMID 30472318
- [Result] Curtin KB, Cheng YI, Wang J, Scott RK, Squires L, Benator DA, Lyon ME; Palliative Care Consortiums. Quality of life of persons living with HIV and congruence with surrogate decision-makers. Qual Life Res. 2019 Jan;28(1):47-56. doi: 10.1007/s11136-018-2002-5. Epub 2018 Sep 15. PMID 30219937
- [Result] Lyon ME, Squires L, Scott RK, Benator D, Briggs L, Greenberg I, D'Angelo LJ, Cheng YI, Wang J. Effect of FAmily CEntered (FACE(R)) Advance Care Planning on Longitudinal Congruence in End-of-Life Treatment Preferences: A Randomized Clinical Trial. AIDS Behav. 2020 Dec;24(12):3359-3375. doi: 10.1007/s10461-020-02909-y. PMID 32399799
- [Result] Grill KB, Wang J, Cheng YI, Lyon ME. The Role of Religiousness and Spirituality in Health-related Quality of Life of Persons Living with HIV: A Latent Class Analysis. Psycholog Relig Spiritual. 2020 Nov;12(4):494-504. doi: 10.1037/rel0000301. Epub 2020 Jan 30. PMID 33777311